CLINICAL TRIAL: NCT00170625
Title: Multicenter, Prospective Phase-I/II-study: Topotecan and Carboplatin in the Therapy of Patients With Relapsed Ovarian Cancer
Brief Title: Therapy With Topotecan and Carboplatin by Patients With Relapsed Ovarian Cancer
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: North Eastern German Society of Gynaecological Oncology (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: NOGGO ov7
Record Dates: First submitted 2005-09-09; First posted 2005-09-15 (Estimated); Results first posted 2017-02-06 (Estimated); Last update posted 2024-11-12 (Actual); Status verified 2024-11

CONDITIONS: Ovarian Cancer
Keywords: platin-resistant
MeSH Terms: conditions — Ovarian Neoplasms | interventions — Topotecan

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Relapse 6-12 months (Experimental): dose level 0: Topotecan 1mg/m2/d on day 1-3, q 21d (+ Carboplatin AUC 5 on day 3 after Topotecan application)
  If dose limiting toxicity (DLT) is present then Topotecan dose will be reduced to dose level -1 (dose level -1: Topotecan 0.75 mg/m2/d on day 1-3, q 21d (+ Carboplatin AUC 5 on day 3 after Topotecan application))
  A DLT is present if a patient has a postponement due to hematologic toxicity of more than 7 days within the first four courses at dose level 0.
  Interventions: Drug: Hycamtin
- Relapse >12 months (Experimental): dose level 0: Topotecan 1mg/m2/d on day 1-3, q 21d (+ Carboplatin AUC 5 on day 3 after Topotecan application)
  If dose limiting toxicity (DLT) is present then Topotecan dose will be reduced to dose level -1 (dose level -1: Topotecan 0.75 mg/m2/d on day 1-3, q 21d (+ Carboplatin AUC 5 on day 3 after Topotecan application))
  A DLT is present if a patient has a postponement due to hematologic toxicity of more than 7 days within the first four courses at dose level 0.
  Interventions: Drug: Hycamtin

INTERVENTIONS:
Drug: Hycamtin — Topotecan: 1,0 mg/m²/d, day 1-3; q21d Carboplatin: AUC 5 on day 3 after Topotecan, q21d

SUMMARY:
Compatibility of the topotecan therapy in combination with carboplatin.

DETAILED DESCRIPTION:
The aim of the study was to confirm the tolerability of 3-day topotecan therapy in combination with carboplatin in accordance with published data and to investigate the tolerability of continued therapy until disease progression or up to a maximum of 12 months.

ELIGIBILITY:
Inclusion Criteria:

* Age >= 18 years
* patient with ovarian cancer after primary therapy
* bone marrow function leukocytes >= 4,0 x 109/ l, platelets >= 100 109/l, hemoglobin >= 9 g/dl
* renal function creatinin <= 1,5 mg% or creatinin clearance >= 60 ml/min
* liver function bilirubin <= 2,0 mg/dl, SGOT, SGPT and AP within 3 fold of the reference laboratory's normal range
* ECOG <= 2
* Intention of regular follow-up visits for the duration of the study
* written informed consent

Exclusion Criteria:

* any known hypersensitivity against topotecan isomerase-I-inhibitor other medication included in the study protocol
* ECOG > 2
* patients with radiotherapy within the last 4 weeks

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 28 (Actual)
Dates: Start 2004-06; Primary Completion 2005-08 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Jalid Sehouli, Principal Investigator — Charite University, Berlin, Germany

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Fotopoulou C, Karavas A, Trappe R, Chekerov R, Lichtenegger W, Sehouli J. Venous thromboembolism in recurrent ovarian cancer-patients: A systematic evaluation of the North-Eastern German Society of Gynaecologic Oncology Ovarian Cancer Study Group (NOGGO). Thromb Res. 2009 Nov;124(5):531-5. doi: 10.1016/j.thromres.2009.03.013. Epub 2009 May 8. PMID 19427025

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Recruitment period: 2.6.2004 - 30.8.2005
Pre-assignment Details: 2 patients missed the inclusion criteria
Period: Overall Study
Arm/Group | Relapse 6-12 Months | Relapse >12 Months
Started | 13 | 13
Completed | 13 | 13
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Relapse 6-12 Months | Relapse >12 Months | Total
Number analyzed (Participants) | 13 | 13 | 26
Age, Continuous [Median (Full Range); unit: years] | 60 [35 to 75] | 63 [28 to 71] | 61.5 [28 to 75]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 13 | 13 | 26
  Male | 0 | 0 | 0
Region of Enrollment [Number; unit: participants]
  Germany | 13 | 13 | 26
Classification of tumour (according to FIGO ovarian cancer staging) [Count of Participants; unit: Participants] — IA - Tumor limited to one ovary, IB - Tumor limited to both ovaries, IC - Tumor involves 1 or both ovaries + capsule rupture, tumor on surface or positive washings/ascites, IIA - Extension and/or implants on the uterus and/or tube(s), IIB - Extension to other pelvic intraperitoneal tissues, IIC - IIA or IIB with positive washings/ascites, IIIA - Microscopic peritoneal metastasis beyond the pelvis, IIIB - Macroscopic, extrapelvic, peritoneal metastasis ≤ 2 cm, IIIC - Macroscopic, extrapelvic, peritoneal metastasis > 2 cm and/or regional lymph node metastasis, IV - Distant metastasis
  Participants
    stage IA | 0 | 1 | 1
    stage IB | 0 | 0 | 0
    stage IC | 0 | 2 | 2
    stage IIA | 0 | 0 | 0
    stage IIB | 0 | 0 | 0
    stage IIC | 1 | 1 | 2
    stage IIIA | 0 | 0 | 0
    stage IIIB | 2 | 0 | 2
    stage IIIC | 8 | 8 | 16
    stage IV | 2 | 1 | 3

OUTCOME MEASURES:

1. Primary Outcome: Occurrence of a DLT (Dose Limiting Toxicity)
Description: A DLT is present if a patient has a postponement due to hematologic toxicity of more than 7 days within the first four courses at dose level 0.
Time Frame: after each cycle for up to one year
Measure: Count of Participants; unit: Participants
Arm/Group | Relapse 6-12 Months | Relapse >12 Months
Number analyzed (Participants) | 13 | 13
Participants | 0 | 1

2. Secondary Outcome: Progression-free Survival (PFS)
Description: Progression-free survival according to kaplan-meier-estimator
Time Frame: after every third cycle, for up to one year
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Relapse 6-12 Months | Relapse >12 Months
Number analyzed (Participants) | 13 | 13
months | 7.3 [1.3 to 14.0] | 8.4 [1.9 to 18.1]

ADVERSE EVENTS:
Time Frame: Until 6 months after 4th study cycle
Description: At each visits patients were asked for the occurence of adverse events and blood samples for laboratory assessment were taken in addition.
Groups:
- Relapse>12 Months: dose level 0: Topotecan 1mg/m2/d on day 1-3, q 21d (+ Carboplatin AUC 5 on day 3 after Topotecan application)
  If dose limiting toxicity (DLT) is present then Topotecan dose will be reduced to dose level -1 (dose level -1: Topotecan 0.75 mg/m2/d on day 1-3, q 21d (+ Carboplatin AUC 5 on day 3 after Topotecan application))
  A DLT is present if a patient has a postponement due to hematologic toxicity of more than 7 days within the first four courses at dose level 0.
Arm/Group | Relapse 6-12 Months | Relapse>12 Months
All-Cause Mortality (participants affected / at risk) | 4/13 | 4/13
Serious Adverse Events (participants affected / at risk) | 6/13 | 6/13
Other Adverse Events (participants affected / at risk) | 10/13 | 7/13
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Relapse 6-12 Months (N=13) | Relapse>12 Months (N=13)
allergic reaction (Immune system disorders) | 0 | 1
anemia (Blood and lymphatic system disorders) | 2 | 1
Thrombocytopenia (Blood and lymphatic system disorders) | 4 | 4
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Relapse 6-12 Months (N=13) | Relapse>12 Months (N=13)
abdominal pain (Gastrointestinal disorders) | 4 | 2
Diarrhea (Gastrointestinal disorders) | 0 | 2
Emesis (Gastrointestinal disorders) | 1 | 1
Constipation (Gastrointestinal disorders) | 3 | 0
Nausea (Gastrointestinal disorders) | 2 | 2

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of more than 60 days